CLINICAL TRIAL: NCT07225283
Title: Developing Resiliency and Exercise Using AI-based Messaging: The DREAM Pilot Study
Brief Title: Developing Resiliency and Exercise Using AI-based Messaging
Acronym: DREAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Celano, Associate Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025P002706
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DREAM (Experimental): Participants will engage in twice weekly, interactive messaging sessions with DREAM, a computer-based messaging system designed to help people engage in more physical activity and improve overall well-being. In the first session of each week, participants will set a physical activity goal and learn a new positive psychology topic. They will review goals and topics from the prior week. In the second session, participants will be reminded of the goals set during the first messaging session earlier that week. The program will run for eight weeks.
  Interventions: Behavioral: DREAM
- Wait-list control (No Intervention): Participants in the wait-list control condition will engage in usual medical care for eight weeks, then will complete the DREAM program.

INTERVENTIONS:
Behavioral: DREAM — Participants will engage in twice weekly messaging sessions and will work towards a physical activity goal each week for a total of eight weeks.
  Arms: DREAM

SUMMARY:
This is a randomized, controlled pilot trial to examine the feasibility, acceptability, and preliminary efficacy of the DREAM program, an 8-week message-based intervention to promote physical activity and well-being in adults with type 2 diabetes.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot trial to examine the feasibility, acceptability, and preliminary efficacy of the DREAM program. DREAM is an 8-week message-based program to promote physical activity and well-being in adults with type 2 diabetes. In DREAM, participants will complete twice weekly messaging sessions, in which they will set weekly physical activity goals and perform activities to enhance well-being. The primary outcome is feasibility (measured by number of messaging sessions successfully transmitted) and acceptability (measured by 0-10 utility ratings). Secondary outcomes include preliminary impact on physical activity and psychological and health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosis (A1c ≥6.5%, fasting glucose ≥126 mg/dL)
* Suboptimal physical activity (score < 5 on the Medical Outcomes Study Specific Adherence Scale physical activity item)
* Access to a smartphone (i.e., Android or iOS) or computer with access to the internet and an internet browser

Exclusion Criteria:

* An unrelated condition limiting physical activity
* Participation in any other programs focused on physical activity or well-being
* A cognitive disturbance precluding participation or informed consent
* Current pregnancy or plan to become pregnant in the next 16 weeks
* Inability to speak/write fluently in English
* Use of non-basal insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delivery of messaging sessions (feasibility) | Twice weekly over 8 weeks
  Proportion of messaging sessions successfully initiated

SECONDARY OUTCOMES:
Utility of the DREAM program | 8 weeks
  Participants will rate the utility of the DREAM program on an 11-point Likert scale (0-10), with 0 being not at all helpful and 10 being very helpful.
Utility of messaging sessions | 8 weeks
  Participants will rate the utility of the messaging sessions, measured on an 11-point Likert scale (0-10), with 0 being not at all helpful and 10 being very helpful.
Change in overall physical activity (in steps/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  Physical activity (steps) will be measured via an Actigraph accelerometer. We will use established accelerometer protocols to measure the mean number of steps taken per day at each time point.
Change in moderate to vigorous physical activity (MVPA; in mean minutes/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  MVPA (reported in mean minutes of MVPA/day) will be measured via an Actigraph accelerometer and recorded in mean minutes/day
Change in positive affect (Positive and Negative Affect Schedule [PANAS] positive affect items) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Positive affect (our main psychological outcome given its links to health outcomes and sensitivity to change) will be assessed via the Positive and Negative Affect Schedule (PANAS) positive affect items. PANAS scores range from 10-50, with higher scores indicating higher levels of positive affect.

OTHER OUTCOMES:
Change in sedentary time (in mean minutes/day) | Measured for 7 days at baseline (both groups), 8-weeks (both groups), and 16 weeks (wait-list control group only)
  Sedentary time (mean minutes/day) will be measured via Actigraph accelerometer.
Change in self-reported physical activity (International Physical Activity Questionnaire [IPAQ]; in metabolic equivalent-minutes/week) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  This will be measured via the International Physical Activity Questionnaire (IPAQ) as a secondary measure of physical activity.
Change in optimism (Life Orientation Test - Revised [LOT-R]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Optimism will be measured using the Life Orientation Test - Revised (LOT-R), a frequently used 6-item instrument that assesses dispositional optimism. LOT-R scores range from 0-24, with higher scores indicating higher levels of optimism.
Change in depressive symptoms (depression subscale of the Hospital Anxiety and Depression Scale [HADS]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Depressive symptoms will be measured using the 7-item depression subscale of the Hospital Anxiety and Depression Scale (HADS). The depression subscale of the HADS ranges from 0-21, with higher scores indicating higher levels of depression.
Change in anxiety (anxiety subscale of the Hospital Anxiety and Depression Scale [HADS]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Anxiety will be measured using the 7-item anxiety subscale of the Hospital Anxiety and Depression Scale (HADS). The anxiety subscale of the HADS ranges from 0-21, with higher scores indicating higher levels of anxiety.
Change in exercise self-efficacy (Self-Efficacy for Exercise scale [SEE]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Exercise self-efficacy will be measured via the Self-Efficacy for Exercise (SEE) scale. SEE scores range from 0-90, with higher scores indicating higher levels of self-efficacy for exercise.
Change in perceived social support (Multidimensional Scale of Perceived Social Support) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Perceived social support will be measured by the Multidimensional Scale of Perceived Social Support (MSPSS). MSPSS scores range from 1-7, with higher scores indicating higher levels of perceived social support.
Change in locus of control (Form C of the Multidimensional Health Locus of Control scale [MHLC Form C]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Locus of control will be measured using the 18-item Multidimensional Health Locus of Control scale [MHLC Form C]. Scores on this scale range from 6-36, with higher scores indicating greater internal health locus of control.
Change in positive affect during activity (Physical Activity Enjoyment Scale) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Positive affect during activity will be measured using the Physical Activity Enjoyment Scale. Physical Activity Enjoyment Scale scores range from 18-126, with higher scores indicating higher levels of enjoyment during activity.
Change in physical health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] physical component score) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  The SF-12 physical component score will be used to assess physical health-related quality of life (Range: 0-100). Higher scores indicate higher levels of physical health-related quality of life.
Change in mental health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] mental component score) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  The SF-12 mental component score will be used to assess mental health-related quality of life (Range: 0-100). Higher scores indicate higher levels of mental health-related quality of life.
Change in adherence to a diabetes diet (General diet items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline (both groups), 8 weeks (both groups), 16 weeks (wait-list control group)
  Measured by the general diet items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate greater adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No